CLINICAL TRIAL: NCT05463003
Title: Impact of OCT1 and CYP2D6 Genotypes on Pharmacokinetics of Berberine in Healthy Volunteers
Acronym: BERKI-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Stefan Engeli, MD, Prof. Dr. med Stefan Engeli, University Medicine Greifswald
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPHA-2022-002
Record Dates: First submitted 2022-07-08; First posted 2022-07-18 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Pharmacokinetic Study in Healthy Volunteers
Keywords: Berberine; OCT1; CYP2D6; pharmacogenetic; pharmacokinetic
MeSH Terms: interventions — Berberine

STUDY DESIGN:
Intervention Model Description: This study should investigate the differences of berberine pharmacokinetic parameters in three cohorts of healthy volunteers:
  Cohort 1a) OCT1 and CYP2D6 wildtype genotypes n = 10 Cohort 1b) OCT1 and CYP2D6 wildtype genotypes n = 10 Cohort 2) OCT1 deficient/CYP2D6 wildtype genotypes n = 10 Cohort 3) OCT1 wildtype/CYP2D6 deficient genotypes n = 10
Masking Description: This Study will be an open label study. Participants will be selected from an existing database of our Institute and are specifically invited according to genotype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OCT1 and CYP2D6 wildtype genotypes (Active Comparator): In this group, the participants are OCT1 and CYP2D6 wildtype genotypes. The participants are selected to achieve best matching according to sex, age, BMI, alcohol consumption and smoking between arm (cohort) 1 and arm (cohort) 2 and 3, respectively.
  Interventions: Dietary Supplement: Berberine
- OCT1 deficient and CYP2D6 wildtype genotypes (Active Comparator): In this group, the participants are OCT1 deficient and CYP2D6 wildtype genotype.
  Interventions: Dietary Supplement: Berberine
- OCT1 wildtype and CYP2D6 deficient genotypes (Active Comparator): In this group, the participants are OCT1 wildtype and CYP2D6 deficient genotype.
  Interventions: Dietary Supplement: Berberine

INTERVENTIONS:
Dietary Supplement: Berberine — A single dose of 1000 mg berberine in two capsules will be administered with 250 ml of still water in the overnight fasting condition. A total of 12 blood samples will be taken at defined time points (baseline, 1; 1.5; 2; 3; 4; 5; 6; 8; 10; 24; 48 h). At each time point, blood will be collected in 2x 7.5 ml tubes for collecting serum and plasma samples to determine berberine, its metabolites and biomarkers of OCT1 transport and CYP2D6 enzymatic activity

SUMMARY:
This study should investigate the differences of berberine pharmacokinetic parameters in three cohorts of healthy volunteers with distinct genotypes of the organic cation transporter 1 (OCT1) gene and the cytochrome P450 2D6 (CYP2D6) gene:

Cohort 1a) OCT1 and CYP2D6 wildtype genotypes n = 10 Cohort 1b) OCT1 and CYP2D6 wildtype genotypes n = 10 Cohort 2) OCT1 deficient/CYP2D6 wildtype genotypes n = 10 Cohort 3) OCT1 wildtype/CYP2D6 deficient genotypes n = 10 Participants will be selected from the study volunteers database of the Institute of Pharmacology in Greifswald according to their OCT1 and CYP2D6 genotypes and to achieve best matching according to sex, age, BMI, alcohol consumption and smoking between Cohort 1a and 2 or Cohort 1b and 3, respectively.

DETAILED DESCRIPTION:
A single dose of 1000 mg berberine will be administered in two capsules with 250 ml of still water in the overnight fasting condition. A total of 12 blood samples will be taken at defined time points (baseline, 1; 1.5; 2; 3; 4; 5; 6; 8; 10; 24; 48 h). At each time point, blood will be collected in 2x 7.5 ml tubes for collecting serum and plasma samples to determine berberine, its metabolites and biomarkers of OCT1 transport and CYP2D6 enzymatic activity. At baseline, additional 2x 2.7 ml blood tubes will be collected for DNA isolation.

The total amount of blood collected for each participant is 190 ml at the three Pharmacokinetic Visits and 10 ml at the Screening Visit. Every hour, participants will drink 100 ml of sparkling water to stimulate intestinal peristalsis and promote transport of the capsule. After 2 hours, the participants may drink a cup of tea or coffee and after 4 hours they will be served a meal. Urine will be collected during the first 10 h after administration. Monitoring of vital parameters, e.g. blood pressure and heart rate, will take place for the first 4 hours after administration. The participants will stay in the Clinical Research Unit of the Institute of Pharmacology for the first 10 hours after administration.

ELIGIBILITY:
Inclusion Criteria:

* any sex
* OCT1 wildtype: homozygous for OCT*1
* OCT "poor transporter": homozygous or heterozygous for OCT1*3, *4, *5, *6
* CYP2D6 wildtype: homozygous or heterozygous for *1, *2, *35
* CYP2D6 "poor metabolizer": homozygous or heterozygous for *3, *4, *5, *6
* age between 18 and 50 years
* understands the study purpose and design
* contractually capable and provides signed informed consent form
* healthy condition or mild and/or well treated forms of allergies, asthma, hypertension, and orthopedic diseases
* a maximum of 3 chronically taken drugs not interfering with OCT1 and CYP2D6 activities

Exclusion Criteria:

* BMI > 35 kg/m2 and <18 kg/m2
* known pregnancy or lactation period
* women: positive urine pregnancy test at screening or pharmacokinetic visit
* anemia (hemoglobin < 13 g/dl (8,07 mmol/l) in men or < 12 g/dl (7,45 mmol/l) in women
* elevated liver function tests (> 2x ULN)
* reduced renal function (eGFRMDRD < 60 ml/min/1,7m2)
* psychiatric disease or drug dependency at time of visit
* use of recreational drugs more than twice a week
* poor venous conditions that make it impossible to place a peripheral venous catheter and regularly draw blood through it

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Berberine plasma and serum concentration expressed as Area under the Curve (AUC0-48 hours). | 48 hours
  Difference in berberine plasma and serum concentrations expressed as Area under the Curve (AUC0-48 hours) between 1) OCT1 wildtype and OCT1 loss of function cohorts (Cohort 1a vs. Cohort 2), and 2) between CYP2D6 wildtype and CYP2D6 loss of function cohorts (Cohort 1b vs. Cohort 3).

SECONDARY OUTCOMES:
Highest concentration (Cmax) of berberine and the berberine metabolites M1-M9. | 48 hours
  Differences in Cmax of berberine and the berberine metabolites M1-M9 between the above described cohorts.
Time point of highest concentration (Tmax) of berberine and the berberine metabolites M1-M9. | 48 hours
  Differences in Tmax of berberine and the berberine metabolites M1-M9 between the above described cohorts.
Clearance of berberine and the berberine metabolites M1-M9. | 48 hours
  Differences in Clearance of berberine and the berberine metabolites M1-M9 between the above described cohorts.
Apparent volume of distribution of berberine and the berberine metabolites M1-M9. | 48 hours
  Differences in apparent volume of distribution of berberine and the berberine metabolites M1-M9 between the above described cohorts.
Changes of plasma concentrations of known endogenous biomarkers like isobutyrylcarnitine | 48 hours
  Changes of plasma concentrations of known endogenous biomarkers like isobutyrylcarnitine. These will be monitored during all time points after berberine administration and their changes over time will be related to the concentration changes of berberine and its major metabolites over time.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Engeli, Prof., Principal Investigator — Universitätsmedizin Greifswald, Institut für Pharmakologie
Locations (1):
- University Medicine Greifswald, Institute of Pharmacology, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blocher JA, Meyer-Tonnies MJ, Morof F, Ronnpagel V, Bethmann J, Vollmer M, Engeli S, Tzvetkov MV. Sex-Dependent Effects of CYP2D6 on the Pharmacokinetics of Berberine in Humans. Clin Pharmacol Ther. 2025 Jan;117(1):250-260. doi: 10.1002/cpt.3454. Epub 2024 Nov 3. PMID 39488825